CLINICAL TRIAL: NCT06617299
Title: Cognitive-Behavioral Intervention Targeting Mothers to Increase Practice of Responsive Feeding and Maintain Healthy Weight in Infants Minors
Brief Title: Cognitive-behavioral Intervention to Increase the Practice of Responsive Feeding and Maintain Healthy Weight in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Collaborators: Universidad de la Sabana (Other)
Responsible Party: Principal Investigator, Jorge Alberto Mayo Abarca, Master in Nursing, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FAEN-D-2017
Record Dates: First submitted 2024-09-24; First posted 2024-09-27 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Prevention Childhood Obesity
Keywords: Infants; Responsive Feeding

STUDY DESIGN:
Intervention Model Description: The present study will be a phase II intervention study of the pilot clinical trial type because the preliminary effect of an intervention will be evaluated where the Experimental Group (EG) will receive the intervention aimed at increasing the practice of RP and maintaining a healthy weight. The Control Group (CG) will receive the usual care, there will be randomization to both groups through a list with the number of rooms, the pilot clinical trial will be of repeated measurements by virtue of which measurements will be made at three times: before the intervention (baseline) and follow-up (post-test 3 and 6 months later) (Grove, Burns & Gray, 2015).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Responsive Feeding Group (Experimental): Group to receive information on responsive feeding
  Interventions: Behavioral: Intervention Identifies and Responds
- Breastfeeding Group (No Intervention): Group to receive information disseminated by hospital staff on breastfeeding

INTERVENTIONS:
Behavioral: Intervention Identifies and Responds — The treatment of Experimental Group is described, which is made up of eight individual sessions taught over three months. Session one will be in face-to-face format, the content, resources and activities are described in tables 2 and 3. The remaining seven sessions will be follow-up sessions (four sessions by message (WhatsApp®) where motivational messages and reinforcement information will be sent; and 3 sessions by phone call for feedback, see details of time, content, activities and resources in tables 2 and 3.
  The design of the intervention is aimed at increasing the practice of Responsive Feeding in mothers with children under 6 months of age, is based on the methodology of Sidani and Braden (2021); on CHW (Bandura, 1986); and behavior change techniques to help people have healthy eating habits (Michie et al., 2011).
  Arms: Responsive Feeding Group

SUMMARY:
Introduction: Childhood overweight and obesity in Mexico is a serious public health problem. Perceptive eating is a factor in the prevention of obesity and occurs when the caregiver recognizes the signs of hunger and satiety, responds in a timely manner to these needs. However, its implementation is often a challenge for parents. Studies show that there is low knowledge and self-efficacy, as well as erroneous beliefs about food. Teaching perceptive eating can lead to: the development of healthy eating habits, generate warm environments in which the interaction between parents and children is strengthened and promote self-regulation of hunger and satiety sensations and prevent overweight and obesity. Interventions on Responsive Feeding for the prevention of healthy weight in infants under six months of age are null in Mexico. Objective: To evaluate the effect of the intervention: "Identify and Respond" aimed at Mexican mothers to increase the practice of Responsive Feeding and maintain a healthy weight in children under 6 months of age. Methodology: The present study will be a pilot clinical trial type intervention study because the preliminary effect will be evaluated where the Experimental Group will receive the intervention aimed at increasing the practice of Responsive Feeding , there will be randomization of repeated measurements by virtue of which measurements will be made at three times: before the intervention (baseline) and follow-up (post-test 3 and 6 months later). The sample consisted of 72 mothers with children younger than 6 months for each group (N=144).

ELIGIBILITY:
Inclusion Criteria:

* Mother/child dyad, apparently healthy.
* Minimum of 12 hours postpartum and/or cesarean section.
* Mother who knows how to read and write.
* Mother who has a smartphone.
* Mother with internet access.
* Mother who agrees to participate in the study.

Exclusion Criteria:

* Hospital stay of the mother/child dyad for more than 7 days after birth.
* Child-related exclusions:
* Gestational age under 37 weeks (SDG).
* Presence of a congenital anomaly.
* Physical disability that could affect feeding (e.g., cleft palate, cleft lip).
* Low birth weight (< 2,500 g).

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Change the practice of responsive feeding in mothers with infants under 6 months of age. | Three measurements will be taken: before the behavioral intervention, 3 months after the intervention and 6 months after the intervention.
  To measure the practice of Responsive Feeding in the mother/child dyad, the Feeding Practices and Structure Questionnaire (FPSQ) will be used, a questionnaire in original English designed by Jansen et al., (2022), replicated in the Mexican context (Pérez, 2023). It aims to measure the responsiveness of parents in children under 6 months, mainly breastfed or bottle-fed throughout childhood. It is made up of 18 items divided into 4 dimensions: 1) on-demand feeding, which refers to the fact that the parents make the decision about when the child should be fed; 2) use of food to calm conceptualized as the fact that parents use food to calm or control emotions; 3) persuasive feeding is the fact that parents encourage (pressure) the child to eat more, even when they show signs of satiety; and 4) parent-directed feeding referring to the fact that the parents make the decision (or have a rule) about how long / how much the child feeds.
Healthy weight maintenance in infants | Three measurements will be taken: before the behavioral intervention, 3 months after the intervention and 6 months after the intervention.
  The nutritional status of the infant will be analyzed through the indicators of weight/length and BMI/age during birth and follow-up measurements, this according to the WHO and the open-access computer program Anthro®, the patterns of child growth in children under two years of age classified by the z-scores will be used : malnutrition (≤ -2 SD); normal (≥ -1 and ≤ 1 SD); SP (> 1 and ≤ 2 DE) and OB (≥ 2 DE).

SECONDARY OUTCOMES:
Mother's Knowledge on the development and feeding practices of the child | Three measurements will be taken: before the behavioral intervention, 3 months after the intervention and 6 months after the intervention.
  To measure the knowledge variable about Responsive Feeding, it will be measured with the Infant Hunger and Satiety Signals Knowledge Scale, originally a scale used in the United States, it was adapted by Ortiz et al. (2020) to the Mexican context, it aims to measure the mother's knowledge regarding the hunger and satiety signals emitted by the infant under 6 months of age. It is structured by 2 questions: 1) Do you know that your child is hungry? with 10 signs to identify them; 2) Do you know that your child is full or full? followed by 8 satiety signals to identify them.
Maternal attitudes Mother's disposition towards infant feeding methods | Three measurements will be taken: before the behavioral intervention, 3 months after the intervention and 6 months after the intervention.
  To measure attitudes towards feeding, the Iowa Infant Feeding Attitude Scale (De la Mora et al., 1999) adapted to the Mexican context by Aguilar-Navarro et al. (2016) will be used, it is a one-dimensional scale made up of 17 items that measure the attitude of mothers towards infant feeding (breastfeeding and/or formula feeding). The way to respond is through a five-point Likert-type scale, where 1) totally disagree; 2) disagree; 3) neither disagree nor agree; 4) agree; 5) Totally agree. It is interpreted that the lower the score, the breastfeeding method is favored and the higher the score, the better attitudes towards formula feeding.
Infant temperament | Three measurements will be taken: before the behavioral intervention, 3 months after the intervention and 6 months after the intervention.
  To measure infant temperament, the Infant Behavior Questionnaire (IBQ-R) (Putnam, 2014) will be used, adapted to the Mexican context by Ortega et al. (2012), its main objective is to measure infant temperament during the last week prior to its application. It is structured by 37 items divided into three dimensions: 1) extroversion; 2) negative affectivity; and 3) self-regulation.
  It has a 7-point Likert-type response scale ranging from 1 = never to 7 = always, for interpretation item 11 evaluates inversely, a sum of the total of the items is made and it is considered that, the higher the score, the greater the characteristic of child temperament according to the three dimensions of the questionnaire.
Parental Self-Efficacy | Three measurements will be taken: before the behavioral intervention, 3 months after the intervention and 6 months after the intervention.
  To measure parental self-efficacy , the Karitane Parental Trust Scale (KPCS) proposed by Crncec et al. (2008) will be used, which aims to measure parental self-efficacy in parents of infants aged 0 to 12 months. It is made up of 15 items divided into three dimensions: 1) perceptions of parenting capacity (5, 4, 6, 2, 8, 7, 3 and 11); 2) available parenting support (15, 13, 9, 14, and 12) and 3) perceptions of child development (10 and 1).
  The structure to answer each of the questions is through a Likert-type scale, where 4 possible options are presented: 0=No, almost never, 1= No, not very often, 2= Yes, sometimes, 3= Yes, most of the time. Despite having dimensions, the authors recommend that its evaluation be done in a one-dimensional way. So if the scores range from 0 to 3, higher scores indicate greater parental self-efficacy, therefore, the range of possible scores on the KPCS is from 0 to 45.
Feeding Self-Efficacy | Three measurements will be taken: before the behavioral intervention, 3 months after the intervention and 6 months after the intervention.
  To measure food self-efficacy , the Food Self-Efficacy Scale proposed by Chen et al. (2022) will be used, which aims to measure maternal self-confidence in their ability to meet feeding demands and successfully perform feeding behavior. It is made up of 5 items in a single dimension.
  The structure to answer each of the questions is through a Likert-type scale, where 4 possible options are presented: 1=Strongly disagree, 2= Disagree, 3= Agree, 4= Strongly agree. Scores range from 1 to 4, higher scores indicate greater food self-efficacy, therefore the range of possible scores on this scale is 4 to 20

CONTACTS AND LOCATIONS:
Overall Officials: Velia M Cárdenas Villareal, PhD, Study Director — Universidad Autónoma de Nuevo León - Facultad de Enfermería; Gabriela I Martínez Figueroa, Master, Study Chair — Universidad Autónoma de Nuevo León - Facultad de Enfermería; Gloria Carvajal Carrascal, PhD, Study Chair — Universidad de la Sabana
Locations (1):
- Hospital Universitario Dr. José Eleuterio González, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No
Personal data will not be shared with other researchers for the protection of personal data included in the study ethics. Only general data derived from the research results will be shared.

REFERENCES:
- [Background] Whitfield KC, Ventura AK. Exploration of Responsive Feeding During Breastfeeding Versus Bottle Feeding of Human Milk: A Within-Subject Pilot Study. Breastfeed Med. 2019 Sep;14(7):482-486. doi: 10.1089/bfm.2019.0069. Epub 2019 Jun 12. PMID 31188021
- [Background] Wen LM, Baur LA, Rissel C, Wardle K, Alperstein G, Simpson JM. Early intervention of multiple home visits to prevent childhood obesity in a disadvantaged population: a home-based randomised controlled trial (Healthy Beginnings Trial). BMC Public Health. 2007 May 10;7:76. doi: 10.1186/1471-2458-7-76. PMID 17490492
- [Background] Vilar-Compte M, Perez-Escamilla R, Orta-Aleman D, Cruz-Villalba V, Segura-Perez S, Nyhan K, Richter LM. Impact of baby behaviour on caregiver's infant feeding decisions during the first 6 months of life: A systematic review. Matern Child Nutr. 2022 May;18 Suppl 3(Suppl 3):e13345. doi: 10.1111/mcn.13345. Epub 2022 Apr 1. PMID 35363420
- [Background] Savage JS, Hohman EE, Marini ME, Shelly A, Paul IM, Birch LL. INSIGHT responsive parenting intervention and infant feeding practices: randomized clinical trial. Int J Behav Nutr Phys Act. 2018 Jul 9;15(1):64. doi: 10.1186/s12966-018-0700-6. PMID 29986721
- [Background] Savage JS, Birch LL, Marini M, Anzman-Frasca S, Paul IM. Effect of the INSIGHT Responsive Parenting Intervention on Rapid Infant Weight Gain and Overweight Status at Age 1 Year: A Randomized Clinical Trial. JAMA Pediatr. 2016 Aug 1;170(8):742-9. doi: 10.1001/jamapediatrics.2016.0445. PMID 27271455
- [Background] Ruggiero CF, Hohman EE, Birch LL, Paul IM, Savage JS. INSIGHT responsive parenting intervention effects on child appetite and maternal feeding practices through age 3 years. Appetite. 2021 Apr 1;159:105060. doi: 10.1016/j.appet.2020.105060. Epub 2020 Dec 1. PMID 33276013
- [Background] Rossiter MD, Richard B, Whitfield KC, Mann L, McIsaac JD. Responsive feeding values and practices among families across the Canadian Maritime provinces. Appl Physiol Nutr Metab. 2022 May;47(5):495-501. doi: 10.1139/apnm-2021-0692. Epub 2022 Feb 3. PMID 35113682
- [Background] Redsell SA, Slater V, Rose J, Olander EK, Matvienko-Sikar K. Barriers and enablers to caregivers' responsive feeding behaviour: A systematic review to inform childhood obesity prevention. Obes Rev. 2021 Jul;22(7):e13228. doi: 10.1111/obr.13228. Epub 2021 Mar 29. PMID 33779040
- [Background] Quah PL, Chan YH, Aris IM, Pang WW, Toh JY, Tint MT, Broekman BF, Saw SM, Kwek K, Godfrey KM, Gluckman PD, Chong YS, Meaney MJ, Yap FK, van Dam RM, Lee YS, Chong MF; GUSTO Study Group. Prospective associations of appetitive traits at 3 and 12 months of age with body mass index and weight gain in the first 2 years of life. BMC Pediatr. 2015 Oct 12;15:153. doi: 10.1186/s12887-015-0467-8. PMID 26459321
- [Background] Putnam SP, Helbig AL, Gartstein MA, Rothbart MK, Leerkes E. Development and assessment of short and very short forms of the infant behavior questionnaire-revised. J Pers Assess. 2014;96(4):445-58. doi: 10.1080/00223891.2013.841171. Epub 2013 Nov 9. PMID 24206185
- [Background] Perez-Escamilla R, Segura-Perez S, Hall Moran V. Dietary guidelines for children under 2 years of age in the context of nurturing care. Matern Child Nutr. 2019 Jul;15(3):e12855. doi: 10.1111/mcn.12855. PMID 31240831
- [Background] Paul IM, Williams JS, Anzman-Frasca S, Beiler JS, Makova KD, Marini ME, Hess LB, Rzucidlo SE, Verdiglione N, Mindell JA, Birch LL. The Intervention Nurses Start Infants Growing on Healthy Trajectories (INSIGHT) study. BMC Pediatr. 2014 Jul 18;14:184. doi: 10.1186/1471-2431-14-184. PMID 25037579
- [Background] Paul IM, Savage JS, Anzman SL, Beiler JS, Marini ME, Stokes JL, Birch LL. Preventing obesity during infancy: a pilot study. Obesity (Silver Spring). 2011 Feb;19(2):353-61. doi: 10.1038/oby.2010.182. Epub 2010 Aug 19. PMID 20725058
- [Background] Pallewaththa P, Agampodi SB, Agampodi TC, Siribaddana SH. Knowledge, Attitudes, and Practices of Responsive Feeding in Rural Sri Lanka (A Qualitative Study). Ceylon Med J. 2019 Jun 30;64(2):70-75. doi: 10.4038/cmj.v64i2.8894. PMID 31455070
- [Background] Paca-Palao A, Huayanay-Espinoza CA, Parra DC, Velasquez-Melendez G, Miranda JJ. [Association between exclusive breastfeeding and obesity in children: a cross-sectional study of three Latin American countries]. Gac Sanit. 2021 Mar-Apr;35(2):168-176. doi: 10.1016/j.gaceta.2019.09.002. Epub 2019 Nov 29. Spanish. PMID 31787405
- [Background] Moura IH, Silva AFRD, Rocha ADESH, Lima LHO, Moreira TMM, Silva ARVD. Construction and validation of educational materials for the prevention of metabolic syndrome in adolescents. Rev Lat Am Enfermagem. 2017 Oct 5;25:e2934. doi: 10.1590/1518-8345.2024.2934. PMID 29020125
- [Background] Michie S, Ashford S, Sniehotta FF, Dombrowski SU, Bishop A, French DP. A refined taxonomy of behaviour change techniques to help people change their physical activity and healthy eating behaviours: the CALO-RE taxonomy. Psychol Health. 2011 Nov;26(11):1479-98. doi: 10.1080/08870446.2010.540664. Epub 2011 Jun 28. PMID 21678185
- [Background] Michie S, Yardley L, West R, Patrick K, Greaves F. Developing and Evaluating Digital Interventions to Promote Behavior Change in Health and Health Care: Recommendations Resulting From an International Workshop. J Med Internet Res. 2017 Jun 29;19(6):e232. doi: 10.2196/jmir.7126. PMID 28663162
- [Background] McNally J, Hugh-Jones S, Hetherington MM. "An invisible map" - maternal perceptions of hunger, satiation and 'enough' in the context of baby led and traditional complementary feeding practices. Appetite. 2020 May 1;148:104608. doi: 10.1016/j.appet.2020.104608. Epub 2020 Jan 11. PMID 31935423
- [Background] Liu Y, Kong Y, Li Z, Zhang G, Wang L, Yu G. Relationships between parental responsive feeding and infant appetitive traits: The moderating role of infant temperament. Front Psychol. 2023 Feb 6;14:1115274. doi: 10.3389/fpsyg.2023.1115274. eCollection 2023. PMID 36814664
- [Background] Lavner JA, Stansfield BK, Beach SRH, Brody GH, Birch LL. Sleep SAAF: a responsive parenting intervention to prevent excessive weight gain and obesity among African American infants. BMC Pediatr. 2019 Jul 5;19(1):224. doi: 10.1186/s12887-019-1583-7. PMID 31277694
- [Background] Kim-Herrera EY, Ramirez-Silva I, Rodriguez-Oliveros G, Ortiz-Panozo E, Sanchez-Estrada M, Rivera-Pasquel M, Perez-Escamilla R, Rivera-Dommarco JA. Parental Feeding Styles and Their Association With Complementary Feeding Practices and Growth in Mexican Children. Front Pediatr. 2021 Dec 21;9:786397. doi: 10.3389/fped.2021.786397. eCollection 2021. PMID 34993164
- [Background] Jansen E, Russell CG, Appleton J, Byrne R, Daniels LA, Fowler C, Rossiter C, Mallan KM. The Feeding Practices and Structure Questionnaire: development and validation of age appropriate versions for infants and toddlers. Int J Behav Nutr Phys Act. 2021 Jan 19;18(1):13. doi: 10.1186/s12966-021-01079-x. PMID 33468156
- [Background] Hernandez E, Lavner JA, Moore AM, Stansfield BK, Beach SRH, Smith JJ, Savage JS. Sleep SAAF responsive parenting intervention improves mothers' feeding practices: a randomized controlled trial among African American mother-infant dyads. Int J Behav Nutr Phys Act. 2022 Oct 1;19(1):129. doi: 10.1186/s12966-022-01366-1. PMID 36183135
- [Background] Hennessy M, Heary C, Laws R, van Rhoon L, Toomey E, Wolstenholme H, Byrne M. The effectiveness of health professional-delivered interventions during the first 1000 days to prevent overweight/obesity in children: A systematic review. Obes Rev. 2019 Dec;20(12):1691-1707. doi: 10.1111/obr.12924. Epub 2019 Sep 2. PMID 31478333
- [Background] Haire-Joshu D, Tabak R. Preventing Obesity Across Generations: Evidence for Early Life Intervention. Annu Rev Public Health. 2016;37:253-71. doi: 10.1146/annurev-publhealth-032315-021859. PMID 26989828
- [Background] Galindo-Neto NM, Alexandre ACS, Barros LM, Sa GGM, Carvalho KM, Caetano JA. Creation and validation of an educational video for deaf people about cardiopulmonary resuscitation. Rev Lat Am Enfermagem. 2019 Mar 10;27:e3130. doi: 10.1590/1518-8345.2765.3130. PMID 30916231
- [Background] Feeley N, Cossette S, Cote J, Heon M, Stremler R, Martorella G, Purden M. The importance of piloting an RCT intervention. Can J Nurs Res. 2009 Jun;41(2):85-99. PMID 19650515
- [Background] Fangupo LJ, Heath AL, Williams SM, Somerville MR, Lawrence JA, Gray AR, Taylor BJ, Mills VC, Watson EO, Galland BC, Sayers RM, Hanna MB, Taylor RW. Impact of an early-life intervention on the nutrition behaviors of 2-y-old children: a randomized controlled trial. Am J Clin Nutr. 2015 Sep;102(3):704-12. doi: 10.3945/ajcn.115.111823. Epub 2015 Jul 29. PMID 26224299
- [Background] Fabrizio CS, Lam TH, Hirschmann MR, Stewart SM. A Brief Parenting Intervention to Enhance the Parent-Child Relationship in Hong Kong: Harmony@Home. J Child Fam Stud. 2013 Jul;22(5):603-613. doi: 10.1007/s10826-012-9614-0. PMID 23772172
- [Background] Dattilo AM, Saavedra JM. Nutrition Education: Application of Theory and Strategies during the First 1,000 Days for Healthy Growth. Nestle Nutr Inst Workshop Ser. 2019;92:1-18. doi: 10.1159/000499544. Epub 2019 Nov 28. PMID 31779004
- [Background] Daniels LA, Mallan KM, Nicholson JM, Thorpe K, Nambiar S, Mauch CE, Magarey A. An Early Feeding Practices Intervention for Obesity Prevention. Pediatrics. 2015 Jul;136(1):e40-9. doi: 10.1542/peds.2014-4108. Epub 2015 Jun 8. PMID 26055848
- [Background] Chen TL, Chien LY. Feeding self-efficacy and feeding outcome expectancy mediate the association between maternal depressive symptoms and responsive feeding. Acta Psychol (Amst). 2022 Oct;230:103755. doi: 10.1016/j.actpsy.2022.103755. Epub 2022 Sep 28. PMID 36179509
- [Background] Cardenas-Villarreal VM, Hernandez-Barrera L, Castro-Sifuentes D, Guevara-Valtier MC, Trejo-Valdivia B. Trends in overweight and obesity in children under 24 months of age in Mexico (2012-2020): analysis of four national health surveys. Cad Saude Publica. 2023 Dec 22;39(12):e00046123. doi: 10.1590/0102-311XEN046123. eCollection 2023. PMID 38126557
- [Background] Cardenas Villarreal VM, Ortiz Felix RE, Cortes-Castell E, Miranda Felix PE, Guevara Valtier MC, Rizo-Baeza MM. [Maternal and infant characteristics associated with obesity in infants under one year of age in northern Mexico]. Nutr Hosp. 2018 Oct 5;35(5):1024-1032. doi: 10.20960/nh.1720. Spanish. PMID 30307282
- [Background] Burnett AJ, Jansen E, Appleton J, Rossiter C, Fowler C, Denney-Wilson E, Russell CG. Bidirectional associations between parental feeding practices, infant appetitive traits and infant BMIz: a longitudinal cohort study. Int J Behav Nutr Phys Act. 2022 Dec 15;19(1):153. doi: 10.1186/s12966-022-01392-z. PMID 36517797
- [Background] Black MM, Tofail F, Hodges EA, Bann CM, Hamadani JD, Aktar S, Lutter CK. Rethinking Responsive Feeding: Insights from Bangladesh. Nutrients. 2022 Jul 30;14(15):3156. doi: 10.3390/nu14153156. PMID 35956330
- [Background] Bahorski J, Romano M, McDougal JM, Kiratzis E, Pocchio K, Paek I. Development of an Individualized Responsive Feeding Intervention-Learning Early Infant Feeding Cues: Protocol for a Nonrandomized Study. JMIR Res Protoc. 2023 Feb 28;12:e44329. doi: 10.2196/44329. PMID 36853761
- [Background] Aguilar-Navarro, H. J., Coronado-Castilleja, A., Gómez-Hernández, O. J., &amp;amp; Cobos-Aguilar, H. (2016). Adaptation of the Iowa Infant Feeding Attitude Scale in the Mexican population. Acta pediátrica de México, 37(3), 149-158.
- See also: Ley General de Salud — https://www.diputados.gob.mx/LeyesBiblio/regley/Reg_LGS_MIS.pdf